CLINICAL TRIAL: NCT07139405
Title: A DOUBLE-BLIND, RANDOMIZED, ACTIVE-CONTROLLED, PARALLEL-GROUP, PHASE II TRIAL TO EVALUATE THE SAFETY, TOLERABILITY, AND SUPERIORITY OF TRIGLYTZA® OVER METFORMIN IN PATIENTS WITH INADEQUATE GLYCEMIC CONTROL OVER 24 WEEKS OF TREATMENT
Brief Title: TRIGLYTZA® VERSUS METFORMIN IN OBESE ADULT TYPE 2 DIABETES (T2DM) PATIENTS OVER 24 WEEKS OF TREATMENT
Acronym: RESILIENCE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Myopharm Limited (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MYP-001; IND136121 (Other: FDA)
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes (T2DM)
Keywords: Type 2 Diabetes; Diabetes; Metformin; Myopharm; Valsartan; Celecoxcib
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Valsartan; Tablets; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: Metformin XR Monotherapy (Active Comparator): Metformin extended release, (taken AM), stable dose up to 1000mg daily
  Interventions: Drug: Metformin XR 1000mg
- Arm 2: TriGlytza Low Dose (Experimental): TriGlytza low dose includes 500mg Metformin-XR (taken AM), 100mg Celecoxcib (AM), and 80mg Valsartan (taken PM)
  Interventions: Drug: Valsartan 80mg Tablet; Drug: Celecoxib (Celebrex®) 100mg; Drug: Metformin XR 500 mg
- Arm 3: TriGlytza High Dose (Experimental): TriGlytza high dose includes 1000mg Metformin-XR (taken AM), 200mg Celecoxcib (AM), and160mg Valsartan (taken PM)
  Interventions: Drug: Metformin XR 1000mg; Drug: Valsartan 160mg tablet; Drug: Celecoxib (Celebrex®) 200mg

INTERVENTIONS:
Drug: Metformin XR 1000mg — Arm 1: Metformin XR 1000mg Monotherapy (taken AM)
  Arms: Arm 1: Metformin XR Monotherapy; Arm 3: TriGlytza High Dose
Drug: Valsartan 80mg Tablet — Arm 2: Valsartan 80mg (taken PM)
  Arms: Arm 2: TriGlytza Low Dose
Drug: Valsartan 160mg tablet — Arm 3: Valsartan 160mg (taken PM)
  Arms: Arm 3: TriGlytza High Dose
Drug: Celecoxib (Celebrex®) 100mg — Arm 2: Celecoxib 100mg (taken AM)
  Arms: Arm 2: TriGlytza Low Dose
Drug: Celecoxib (Celebrex®) 200mg — Arm 3: Celecoxib (taken AM)
  Arms: Arm 3: TriGlytza High Dose
Drug: Metformin XR 500 mg — Arm 2: Metformin 500mg (taken AM)
  Arms: Arm 2: TriGlytza Low Dose

SUMMARY:
Type 2 diabetes (T2DM) is still very difficult to treat because current medicines mostly help with symptoms but don't stop the damage happening inside the pancreas. Many people who start on common treatments like Metformin, and even newer drugs like Ozempic, eventually stop responding to them. This is because these drugs don't address the real problem: the gradual loss of the pancreas' ability to make insulin and the body's increasing resistance to it.

Myopharm is developing a new treatment called TriGlytza®, which combines existing medicines (Celecoxib and Valsartan) with Metformin. This new approach is designed to target the inflammation and biological pathways that cause ongoing damage in Type 2 diabetes, aiming to protect the pancreas and reduce insulin resistance. Early animal studies and past clinical trials with the individual drugs show promising results.

The number of people with Type 2 diabetes is expected to double by 2045, and the disease brings huge health and financial costs. It also raises the risk of heart disease, stroke, kidney damage, nerve problems, vision loss, certain cancers, and even conditions like Alzheimer's. Because of this, a treatment that addresses the root causes rather than just symptoms could make a major difference.

TriGlytza® aims to provide a safe, affordable, and more effective long-term treatment than current options, helping people manage their diabetes better and avoid related health problems.

DETAILED DESCRIPTION:
Type 2 diabetes (T2DM) continues to be a major unmet medical need largely due to the currently marketed treatment options not adequately treating the underlying pathophysiology of immune mediated damage to the pancreas.

In real-world clinical practice, first-line therapies with Metformin inadequately control newly diagnosed patients and despite second-line and third-line add-on therapies like Ozempic failure rate continue to be 50% in 2022. These drugs are approved for primarily treating the symptoms of T2DM, Metformin providing short term improvements in insulin sensitivity, and Ozempic stimulating beta cells to make insulin, as indicated by reductions in the HbA1c levels, but not for mitigating the underlying pathophysiology of progressive deterioration of pancreatic beta cell function.

These and other standard prescribed drugs like SGLT2 inhibitors are inadequate in filling one of the most important clinical gaps in the T2DM space: sustained glycemic control via preventing pancreatic beta cell failure and decreasing insulin resistance.

To fill this important gap, Myopharm is developing an innovative patient-centric product: TriGlytza® consisting of Celecoxib, Valsartan treatment add-on to Metformin first-line therapy in diabetes. It is custom-designed to target multiple distinct and overlapping pro-inflammatory signalling pathways along the RAS-IL1b-Cox2-PGE2-EP3 axes that contribute to progressive deterioration of beta cell function and insulin resistance, the core defects observed in T2DM patients. The scientific rationale and the product concept are supported by results obtained from translational animal models of the combination as well as controlled clinical studies with Celecoxib monotherapy and Valsartan monotherapy.

The Type 2 diabetes population is expected to double to over 600 million worldwide by 2045, with the current estimated global economic burden over $2.3 Trillion. The Type 2 diabetes market is expected to be over $58.7B in 2025. The burden of Type 2 diabetes rises substantially with multiple diabetes-related co-morbidities such as coronary artery disease, peripheral arterial disease, stroke, retinopathy, nephropathy, and neuropathy. Additionally, there is 35% increased risk of incidence for cancers such as breast, rectum, pancreas, liver and gall bladder due to T2DM and increased risk of developing Alzheimer's, Parkinson's, and depression in diabetes patients. The link between insulin resistance of the brain cells and Alzheimer's disease is so strong that some have proposed classifying it as Type 3 diabetes.

Unlike the currently marketed treatment options which treat Type 2 diabetes, TriGlytza® is custom designed to treat the disease in the context of these multi-factorial comorbidities and coexisting conditions. This study is designed to show how TriGlytza® is a safe, innovative, and commercially viable superior treatment, differentiated from currently marketed drugs for patients to adequately control their Type 2 diabetes and prevent co-morbidities. TriGlytza® potentially provides an inexpensive and safe option to treat this major unmet medical need.

Results obtained from clinical studies with Type 2 diabetes patients and the translation animal models strongly suggest that TriGlytza® has properties that differentiate it from currently marketed drugs. Its potential to prevent or delay Metformin failure and the observed reduction in risk of insulin dependence in particular warrants evaluation of its superiority over Metformin monotherapy in patients with inadequate glycemic control.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, age 18 and ≤70 at time of screening visit
2. WOCBP must have negative serum or urine pregnancy test (min sensitivity 25 IU/L or equivalent HCG) within 24 hours prior to the start of the study
3. Women must not be breastfeeding
4. Inadequate BG control with Metformin defined as a screening HbA1c of ≥7.0 and ≤ 10.5 at the screening visit
5. Subjects should have been taking the same daily dose of Metformin for at least 8 weeks prior to the enrolment visit and subjects must not receive other antihyperglycemic medications within the 12 weeks prior to screening
6. FPG ≥140 mg/dL
7. BMI ≥28 and ≤40
8. Grade 1 hypertension defined as 140-159 systolic and 90-99 diastolic mmHg if patients is not receiving anti-hypertensive medication at the time of screening / or has never received anti-hypertensive medication.

   If patient is receiving anti-hypertensive medication at the time of screening and their BP is controlled, BP should be within the normal range of <120-139 systolic and <80-89 diastolic.

   Patients receiving anti-hypertensive medication at the time of screening and for which their hypertension is uncontrolled, will be excluded
9. eGFR ≥ 60 ml/min

Exclusion Criteria:

1. Patients with Type 1 Diabetes
2. Patients with history of ketoacidosis
3. Subjects at serious risk of GI adverse events per the discretion of the study site investigator (e.g current or recent history of GI bleeding ulceration, or perforation)
4. Subjects with a planned radiologic study with IV contrast, surgery, or other planned procedures that may predispose them to metformin-associated lactic acidosis
5. Subjects with a history of uncontrolled hyperglycemia (>15.0 mmol/L) after an overnight fast that required rescue therapy
6. Impaired kidney function defined as eGFR ≤60 mL/min
7. Subjects taking any prohibited medications.
8. Any of the following cardiovascular (CV)/vascular diseases within 3 months of the screening visit:

   1. Myocardial infarction (MI)
   2. Cardiac surgery or revascularization (coronary artery bypass surgery, Coronary Artery Bypass Graft [(CABG]/Percutaneous transluminal coronary angioplasty (PTCA)]
   3. Unstable angina
   4. Unstable congestive heart failure (CHF)
   5. Transient ischemic attack (TIA) or significant cerebrovascular disease
   6. Unstable or previously diagnosed arrhythmia
   7. Congestive heart failure, defined as New York Heart Association (NYHA) Class III and IV, unstable or acute heart failure and/or known left ventricular ejection fraction of ≤40%.
   8. Acute coronary syndrome, stroke or transient ischemic attack within 3 months prior to the informed consent
9. Previous bariatric surgery
10. Previous bariatric surgery
11. Treatment with anti-obesity drugs within 3 months prior to screening visit
12. Subjects with COPD
13. Subjects with active liver disease
14. Subjects with active renal disease
15. Subjects with autoimmune diseases e.g. Lupus, Psoriasis
16. Subjects with HIV / AIDS
17. Subjects with Hematological and Oncological Diseases/Conditions
18. Haemoglobin <11.0 g/dL (110 g/L) for men; haemoglobin <10.0 g/dL (100 g/L) for women
19. Subjects with chronic disease e.g. Cancer, Epilepsy, Alzheimer, Parkinson
20. Subjects with abnormal free T4
21. Subjects with serious active infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
To demonstrate that after 24 weeks of treatment, the mean improved change in glycemic response from baseline, measured through mean reduction in HbA1c levels, for TriGlytza™ is superior to Metformin monotherapy. | 24 weeks
  Mean change in HbA1c from baseline to Treatment Week 24.

CONTACTS AND LOCATIONS:
Overall Officials: George Tachas, Study Director — Myopharm Limited

IPD SHARING:
Plan to Share IPD: Undecided
The data will be shared, a plan is being formulated for data sharing and will be uploaded prior to the study activation.